CLINICAL TRIAL: NCT01381666
Title: Evaluation of the Diagnostic Utility of INS316 in Patients With Interstitial Lung Diseases (01-701)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 01-701
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Inhalation; Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- INS316 (Experimental): inhalation via nebulizer given for 2 doses for 60 minutes each
  Interventions: Drug: INS316 solution for inhalation
- hypertonic saline 3% sodium chloride solution (Placebo Comparator): inhalation via nebulizer given for 2 doses for 60 minutes each
  Interventions: Drug: hypertonic saline 3% sodium chloride solution

INTERVENTIONS:
Drug: INS316 solution for inhalation — inhalation via nebulizer given for 2 doses for 60 minutes each
  Arms: INS316
Drug: hypertonic saline 3% sodium chloride solution — inhalation via nebulizer given for 2 doses for 60 minutes each
  Arms: hypertonic saline 3% sodium chloride solution

SUMMARY:
The objective of the present work is to explore and compare the diagnostic quality of sputum specimens obtained by BAL, induction with hypertonic saline (3%), and induction with INS316 in patients diagnosed with interstitial lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* between 18 years or older
* undergone diagnostic bronchoalveolar lavage within the previous 21 days
* diagnosed with sarcoidosis or other ILD

Exclusion Criteria:

* having resting hypoxemia
* receiving corticosteroid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-01; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
diagnosis of sarcoidosis using sputum induction (sputum weight) | 60 minutes

SECONDARY OUTCOMES:
adverse events | 60 minutes